CLINICAL TRIAL: NCT05781243
Title: Normal Saline Versus Lactated Ringer's Solution for Acute Pancreatitis Resuscitation, an Open-label Multicenter Randomized Controlled Trial: the WATERLAND Trial
Brief Title: Normal Saline Versus Lactated Ringer's Solution for Acute Pancreatitis Resuscitation
Acronym: WATERLAND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Enrique de-Madaria (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Universidad Miguel Hernandez de Elche (Other); Hospital del Mar (Other); Hospital Clinico Universitario de Santiago (Other); Hospital Clínico Universitario de Valencia (Other); Hospital Costa del Sol (Other); Corporacion Parc Tauli (Other); Hospital Clínico Universitario Lozano Blesa (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario La Fe (Other); Hospital Miguel Servet (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Universitario Insular Gran Canaria (Other); University Hospital Virgen de las Nieves (Other); Hospital Universitario de Burgos (Other); Hospital Universitario Lucus Augusti (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospital Universitario Puerta del Mar (Other); Instituto de Investigación Sanitaria Hospital Universitario de la Princesa (Other); Dr. Negrin University Hospital (Other); Hospital Regional de Alta Especialidad del Bajio (Other); Asian Institute Of Medical Sciences (Other); Hospital Dr. Jaime Mendoza Sucre Bolivia (Unknown); Hayatabad Medical Complex (Other Government); University Hospital Olomouc (Other); SIDS Hospital & Research Centre Gujarat India (Unknown); Sanatorio Allende (Other); University Hospital Bratislava (Other); University Hospital Sestre Milosrdnice (Other); Attikon Hospital (Other); Nuevo Hospital Iturraspe Santa Fe Argentina (Unknown); Hospital Nacional Rosales (Other); Zagazig University (Other Government); University of Utah (Other); Hospitales Universitarios Virgen del Rocío (Other); University Hospital of Girona Dr. Josep Trueta (Network); Hospital of Navarra (Other); Hospital Clínico Universitario de Valladolid (Other); Hospital Universitario Central de Asturias (Other); Kalinga Hospital, Bhubaneswar (Other); Ohio State University (Other); Zhengzhou University (Other); Jinling Hospital, China (Other); Hospital Privado de Cordoba, Argentina (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other); Postgraduate Institute of Medical Education and Research in Chandigarh (Other); RML Specialty Hospital (Other); Wannan Medical College Yijishan Hospital (Other); Bucharest Emergency Hospital (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other); Emergency County Hospital Pius Brinzeu; Timisoara, Romania (Network); King Hamad University Hospital, Bahrain (Other)
Responsible Party: Sponsor-Investigator, Enrique de-Madaria, Principal Investigator of clinical pancreatology research group-ERICA consortium, ISABIAL, Hospital General Universitario de Alicante
Organization: Hospital General Universitario de Alicante (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eudract 2023-000010-18
Record Dates: First submitted 2023-02-25; First posted 2023-03-23 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Acute Pancreatitis
Keywords: Normal saline; Lactated Ringer solution; Acute pancreatitis; Fluid Therapy; Fluid resuscitation
MeSH Terms: conditions — Pancreatitis | interventions — Ringer's Lactate; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactated Ringer solution (LR) (Experimental): LR: Lactated Ringer solution. Patients in the LR treatment arm will receive fluid therapy based on lactated Ringer's solution for a minimum of 48 hours.
  Interventions: Drug: Lactated Ringer Solution
- Normal saline (NS) (Active Comparator): NS: Normal Saline. Patients in the NS treatment arm will receive fluid therapy based on normal saline for a minimum of 48 hours.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lactated Ringer Solution — Patients in the LR (Lactated Ringer solution) treatment arm will receive fluid therapy based on lactated Ringer's solution for a minimum of 48 hours.
  Arms: Lactated Ringer solution (LR)
Drug: Normal saline — Patients in the NS (Normal Saline) treatment arm will receive fluid therapy based on lactated Ringer's solution for a minimum of 48 hours.
  Arms: Normal saline (NS)

SUMMARY:
Background: Some evidence suggests that fluid resuscitation with lactated Ringer's solution (LR) may have an anti-inflammatory effect on acute pancreatitis (AP) when compared to normal saline (NS), and may be associated with a decrease in severity, but existing single center randomized controlled trials showed conflicting results. The WATERLAND trial aims to investigate the efficacy and safety of fluid resuscitation using LR compared to NS in patients with AP.

Methods: The WATERLAND trial is an international multicenter, open-label, parallel-group, randomized, controlled, superiority trial. Patients will be randomly assigned in a 1:1 ratio to receive LR versus NS-based fluid resuscitation for at least 48 hours. The primary outcome will be moderately severe or severe AP, according to the revision of the Atlanta classification. The secondary objectives of the WATERLAND trial are to determine the effect of LR versus NS fluid resuscitation on several efficacy and safety outcomes in patients with AP.

A total sample of 720 patients, 360 in the LR group and 360 in the NS group, will achieve 90% power to detect a difference between the group proportions of 10%, assuming that the frequency of moderately severe or severe AP in the LR group will be 17%. A loss to follow-up of 10% of patients is expected, so the total sample size will be 396 patients in each treatment arm (792 patients overall). The test statistic used is the two-sided Z test with pooled variance set at a 0.05 significance level.

Discussion: The WATERLAND study aims to improve the early management of AP. Fluid resuscitation is an inexpensive treatment available in any hospital center worldwide. If a better evolution of pancreatitis is demonstrated in one of the treatment arms, it would have important repercussions in the management of this frequent disease.

DETAILED DESCRIPTION:
The entire protocol is published in open-access format, including the Statistical Analysis plan, in the journal Trials: https://doi.org/10.1186/s13063-024-08539-2

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years or older
* Diagnosis of acute pancreatitis according to the revision of the Atlanta classification (Banks et al, Gut 2013), which requires at least two of the following three criteria: A) typical abdominal pain, B) increase in serum amylase or lipase levels higher than three times the upper limit of normality, and C) signs of acute pancreatitis in imaging
* Signature of informed consent

Exclusion Criteria:

* New York Heart Association class II heart failure (slight limitation of physical activity; fatigue, palpitations, or dyspnea with ordinal physical activity) or worse, or ejection fraction <50% in the last echocardiography
* Decompensated cirrhosis (Child's class B or C)
* Hyper or hyponatremia (<135 or >145 mEq/L)
* Hyperkalemia (>5 mEq/L)
* Hypercalcemia (albumin or protein-corrected calcium >10.5 mg/dL or 2.62 mmol/L)
* Criteria for moderately severe or severe acute pancreatitis (revision of the Atlanta classification, Banks et al, Gut 2013) at recruitment: any of the following: A) presence of creatinine ≥1.9 mg/dL or ≥170 mmol/l, B) PaO2/FiO2≤300, C) systolic blood pressure <90 mmHg despite initial fluid resuscitation, D) presence of local complications (acute peripancreatic fluid collections, acute necrotic collection, pseudocyst, walled-off necrosis, gastric outlet dysfunction, splenic or portal vein thrombosis, or colonic necrosis), E) exacerbation of previous comorbidity such as coronary artery disease or chronic lung disease, precipitated by the acute pancreatitis
* Signs of volume overload or heart failure at recruitment (peripheral edema, pulmonary rales, or increased jugular ingurgitation at 45º)
* Time from pain onset to arrival to emergency room >24 h
* Time from confirmation of pancreatitis to randomization >8 h
* Chronic pancreatitis defined by a Wirsung duct ≥4mm and/or pancreatic calcifications
* More than 1 previous episode of acute pancreatitis (only 2 episodes of acute pancreatitis are allowed, one of them the present episode)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with moderately severe or severe acute pancreatitis | From date of randomization until 30 days after randomization
  Presence of local complications, exacerbation of previous comorbidity or organ failure, according to the definitions of these complications provided by the revised Atlanta Classification (https://doi.org/10.1136/gutjnl-2012-302779)

SECONDARY OUTCOMES:
Number of participants with local complications | From date of randomization until 30 days after randomization
  Presence of acute peripancreatic fluid collections, acute necrotic collection, pseudocyst, walled-off necrosis, gastric outlet dysfunction, splenic or portal vein thrombosis, and colonic necrosis according to the revised Atlanta Classification (https://doi.org/10.1136/gutjnl-2012-302779).
Number of participants with necrotizing pancreatitis | From date of randomization until 30 days after randomization
  Presence of acute necrotic collections according to the revised Atlanta Classification (https://doi.org/10.1136/gutjnl-2012-302779).
Number of participants with infection of pancreatic collections or necrosis | From date of randomization until 30 days after randomization
  Extraluminal gas in the pancreatic and/or peripancreatic tissues on CT scan or when a sample from the collection/necrosis contains pus or is positive for bacteria and/or fungi on Gram stain or culture.
Number of participants with systemic inflammatory response syndrome | At 24 and 48 hours
  At least 2 criteria: A) pulse >90 beats/min, B) respirations >20/min or arterial blood PaCO2 <32 mm Hg, C) temperature <36°C or >38°C, D) white blood cell count <4,000 cells/mm3 or >12,000 cells/mm3 or >10% bands
Number of systemic inflammatory response syndrome criteria | At 24 and 48 hours
  The criteria are: A) pulse >90 beats/min, B) respirations >20/min or arterial blood PaCO2 <32 mm Hg, C) temperature <36°C or >38°C, D) white blood cell count <4,000 cells/mm3 or >12,000 cells/mm3 or >10% bands
PAN-PROMISE symptom scale | At 24 and 48 hours (final value and change from baseline)
  PAN-PROMISE scale: a 7-symptom scale patient-reported outcome (range, 0 to 10 for each symptom; overall range, 0 to 70, with higher scores indicating higher symptom intensity). Details: https://doi.org/10.1136/gutjnl-2020-320729
Time to oral refeeding | From date of randomization until 30 days after randomization
  Days from baseline to oral refeeding
Number of participants with invasive treatment | From date of randomization until 30 days after randomization
  Any of the following: thoracocentesis due to pancreatitis-induced pleural effusion, percutaneous and/or endoscopic drainage of pancreatic or peripancreatic fluid collections or necrosis, endoscopic or surgical necrosectomy, endoscopic retrograde cholangiopancreatography due to A) ruptured common bile duct, B) jaundice caused by compression of the common bile duct, C) main pancreatic duct leakage
Number of participants with nutritional support | From date of randomization until 30 days after randomization
  Use of enteral (nasogastric or nasojejunal) or parenteral feeding
Number of participants with intensive care unit admission | From date of randomization until 30 days after randomization
  Admission in the intensive care unit
Number of participants with exacerbation of coexisting condition | From date of randomization until 30 days after randomization
  Exacerbation of pre-existing co-morbidity. The definition provided by the Revised Atlanta Classification is " Exacerbation of pre-existing co-morbidity, such as coronary artery disease or chronic lung disease, precipitated by the acute pancreatitis is defined as a systemic complication. In this document, we distinguish between persistent organ failure (the defining feature of severe acute pancreatitis) and other systemic complications, which are an exacerbation of pre-existing co-morbid disease." (revised Atlanta classification: https://doi.org/10.1136/gutjnl-2012-302779) For the WATERLAND trial we define exacerbation of pre-existing co-morbidity as
Number of participants with any organ failure | From date of randomization until 30 days after randomization
  Definition according to the revised Atlanta classification (https://doi.org/10.1136/gutjnl-2012-302779): organ failure is defined by the presence of any of the following criteria: A) kidney failure as a creatinine ≥1.9 mg/dL or >170 micromol/L, B) cardiovascular failure as a systolic blood pressure <90 mmHg despite fluid resuscitation, and C) respiratory failure as a PaO2/FIO2≤300
Number of participants with persistent organ failure | From date of randomization until 30 days after randomization
  Organ failure lasting more than 48h (revised Atlanta classification: https://doi.org/10.1136/gutjnl-2012-302779)
Number of participants with shock | From date of randomization until 30 days after randomization
  Systolic blood pressure <90 mmHg despite fluid resuscitation (revised Atlanta classification: https://doi.org/10.1136/gutjnl-2012-302779)
Number of participants with respiratory failure | From date of randomization until 30 days after randomization
  PaO2/FIO2≤300 (revised Atlanta classification: https://doi.org/10.1136/gutjnl-2012-302779)
Number of participants with kidney failure | From date of randomization until 30 days after randomization
  Creatinine ≥1.9 mg/dL or >170 micromol/L (revised Atlanta classification: https://doi.org/10.1136/gutjnl-2012-302779)
Mortality (number of participants) | From date of randomization until 30 days after randomization
  Death
Hospital stay | From date of randomization until 30 days after randomization
  Days from recruitment to discharge from index admission
C-reactive protein | At 48 hours from randomization
  C-reactive protein blood levels
Number of participants with hypovolemia | At 24 and 48 hours from randomization
  WATERFALL trial criteria for hypovolemia (see https://www.nejm.org/doi/10.1056/NEJMoa2202884)
Number of participants with fluid overload | From randomization to 72 h thereafter
  WATERFALL trial criteria for fluid overload (see https://www.nejm.org/doi/10.1056/NEJMoa2202884)
Number of participants with acute kidney injury | At 24 and 48 hours from randomization
  KDIGO criteria: increase in serum creatinine of ≥0.3 mg/dL within 48 hr or ≥50% within 7 days or urine output of <0.5 mL/kg/hr for >6 hr (https://doi.org/10.1159/000339789)
Number of participants with hyperkalemia | At 24 and 48 hours from randomization
  Venous potassium>5mEq/L
Number of participants with hypercalcemia | At 24 and 48 hours from randomization
  Venous calcium corrected by proteins>10.5mg/dL or 2.62 mmol/L
Number of participants with hyperchloremia | At 24 and 48 hours from randomization
  Venous chloride>106mEq/L
Number of participants with acidosis | At 24 and 48 hours from randomization
  Venous blood pH <7.35
Number of participants with hyperchloremic acidosis | At 24 and 48 hours from randomization
  Patients with venous chloride>106mEq/L and venous blood pH <7.35
Number of participants with composite safety outcome (primary safety outcome) | At 24 and 48 hours from randomization
  Fluid overload or acute kidney injury or hyperkalemia or hypercalcemia or hyperchloremia or acidosis

CONTACTS AND LOCATIONS:
Overall Officials: Enrique de-Madaria, MD PhD, Principal Investigator — Dr. Balmis General University Hospital
Locations (1):
- Dr. Balmis General University Hospital, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
Members of the ERICA consortium that recruited patients in the WATERLAND trial may claim access to the final dataset to perform post-hoc studies; these proposals will be studied by the steering committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available upon publication of the main study.
Access Criteria: 1. Have enrolled patients in the WATERLAND study.
  2. The Steering Committee will evaluate the project and decide whether it is of sufficient scientific quality.

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] de-Madaria E, Buxbaum JL, Maisonneuve P, Garcia Garcia de Paredes A, Zapater P, Guilabert L, Vaillo-Rocamora A, Rodriguez-Gandia MA, Donate-Ortega J, Lozada-Hernandez EE, Collazo Moreno AJR, Lira-Aguilar A, Llovet LP, Mehta R, Tandel R, Navarro P, Sanchez-Pardo AM, Sanchez-Marin C, Cobreros M, Fernandez-Cabrera I, Casals-Seoane F, Casas Deza D, Lauret-Brana E, Marti-Marques E, Camacho-Montano LM, Ubieto V, Ganuza M, Bolado F; ERICA Consortium. Aggressive or Moderate Fluid Resuscitation in Acute Pancreatitis. N Engl J Med. 2022 Sep 15;387(11):989-1000. doi: 10.1056/NEJMoa2202884. PMID 36103415
- [Background] de-Madaria E, Sanchez-Marin C, Carrillo I, Vege SS, Chooklin S, Bilyak A, Mejuto R, Mauriz V, Hegyi P, Marta K, Kamal A, Lauret-Brana E, Barbu ST, Nunes V, Ruiz-Rebollo ML, Garcia-Rayado G, Lozada-Hernandez EE, Pereira J, Negoi I, Espina S, Hollenbach M, Litvin A, Bolado-Concejo F, Vargas RD, Pascual-Moreno I, Singh VK, Mira JJ. Design and validation of a patient-reported outcome measure scale in acute pancreatitis: the PAN-PROMISE study. Gut. 2021 Jan;70(1):139-147. doi: 10.1136/gutjnl-2020-320729. Epub 2020 Apr 3. PMID 32245906
- [Background] Guilabert L, Cardenas-Jaen K, Vaillo-Rocamora A, Garcia Garcia de Paredes A, Chhoda A, Sheth SG, Lopez-Valero C, Zapater P, Navarrete-Munoz EM, Maisonneuve P, Hernandez-Barco YG, Capurso G, Buxbaum JL, de-Madaria E; ERICA consortium. Normal saline versus lactated Ringer's solution for acute pancreatitis resuscitation, an open-label multicenter randomized controlled trial: the WATERLAND trial study protocol. Trials. 2024 Oct 21;25(1):699. doi: 10.1186/s13063-024-08539-2. PMID 39434191
- See also: Published study protocol and statistical analysis plan — https://pmc.ncbi.nlm.nih.gov/articles/PMC11492666/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/43/NCT05781243/Prot_SAP_000.pdf